CLINICAL TRIAL: NCT02767804
Title: Phase 3 Randomized Study Comparing X-396 (Ensartinib) to Crizotinib in Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: eXalt3: Study Comparing X-396 (Ensartinib) to Crizotinib in ALK Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X396-CLI-301
Record Dates: First submitted 2016-04-30; First posted 2016-05-10 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ALK-positive NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- X-396 (ensartinib) (Experimental): Eligible patients with ALK+ NSCLC will receive oral X-396 (ensartinib) at 225mg QD with or without food until progression or unacceptable toxicity develops
  Interventions: Drug: X-396 (ensartinib)
- crizotinib (Active Comparator): Eligible patients with ALK+ NSCLC will receive oral crizotinib at 250mg BID with or without food until progression or unacceptable toxicity develops
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: X-396 (ensartinib) — oral ALK inhibitor
  Arms: X-396 (ensartinib)
Drug: crizotinib — oral ALK inhibitor
  Other Names: Xalkori
  Arms: crizotinib

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of X-396 (ensartinib) vs. crizotinib in patients with ALK-positive non-small cell lung cancer that have received up to 1 prior chemotherapy regimen and no prior ALK inhibitor.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of X-396 (ensartinib) vs. crizotinib in patients with ALK-positive NSCLC that have received up to 1 prior chemotherapy regimen and no prior ALK tyrosine kinase inhibitor (TKI), to obtain additional pharmacokinetic (PK) data from sparse PK sampling, to compare the quality of life (QoL) in patients receiving X-396 vs. crizotinib, to evaluate the status of exploratory biomarkers and correlate with clinical outcome, and to obtain germline DNA samples for possible pharmacogenetic analysis in the event that outliers with respect to efficacy, tolerability/safety, or exposure are identified.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive by an FDA-approved assay performed centrally. Patients must be ALK positive by local test prior to submitting tissue to the central lab. Randomization will occur after ALK positive confirmation is received from the central lab. Patients may have received up to 1 prior chemotherapy regimen for metastatic disease, which may also include maintenance therapy. Note that patients that have received adjuvant or neoadjuvant chemotherapy and developed metastatic disease within 6 months from the end of that therapy would be considered to have received 1 prior regimen for metastatic disease.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2. (see Appendix A)
3. Life expectancy of at least 12 weeks.
4. Ability to swallow and retain oral medication.
5. Adequate organ system function, defined as follows:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109/L
   2. Platelets ≥100 x 109/L
   3. Hemoglobin ≥9 g/dL (≥90 g/L) Note that transfusions are allowed to meet the required hemoglobin level
   4. Total bilirubin ≤1.5 times the upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN if no liver involvement or ≤5 x ULN with liver involvement.
   6. Creatinine < 1.5 x ULN. If >1.5 x ULN, patient may still be eligible if calculated creatinine clearance >50 mL/min (0.83mL/s) as calculated by the Cockcroft-Gault method.
6. Brain metastases allowed if asymptomatic at study baseline. Patients with untreated brain metastases must not be on corticosteroids. If patients have neurological symptoms or signs due to CNS metastases, patients need to complete whole brain radiation or focal treatment at least 14 days before start of study treatment and be asymptomatic on stable or decreasing doses of corticosteroids at baseline.
7. Men with partners of childbearing potential willing to use adequate contraceptive measures during the study and for 90 days after the last dose of study medication.
8. Women who are not of child-bearing potential, and women of child-bearing potential who agree to use adequate contraceptive measures during the study and for 90 days after the last dose of study medication, and who have a negative serum or urine pregnancy test within 1 week prior to initial trial treatment.
9. Patients must be >18 years-of-age.
10. Patients must have measurable disease per RECIST v. 1.1.
11. Willingness and ability to comply with the trial and follow-up procedures.
12. Ability to understand the nature of this trial and give written informed consent.

Note the following pertains to patients enrolled in France

In France, a subject will be eligible for inclusion in this study only affiliated to the French Social Security system, and currently benefit from the corresponding rights and cover.

Exclusion Criteria

1. Patients that have previously received an ALK TKI or PD-1/PD-L1 therapy, and patients currently receiving cancer therapy (i.e., other targeted therapies, chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
2. Use of an investigational drug within 21 days prior to the first dose of study drug. Note that to be eligible, any drug-related toxicity should have recovered to Grade 1 or less, with the exception of alopecia.
3. Any chemotherapy within 4 weeks, or major surgery or radiotherapy within the last 14 days.
4. Patients with primary CNS tumors and leptomeningeal disease are ineligible.
5. Patients with a previous malignancy within the past 3 years (other than curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, or any cancer that is considered to be cured and have no impact on PFS and OS for the current NSCLC).
6. Concomitant systemic use of anticancer herbal medications. These should be stopped prior to study entry.
7. Patients receiving

   1. strong CYP3A inhibitors (including, but not limited to, atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, grapefruit, grapefruit juice)
   2. strong CYP3A inducers (including, but not limited to, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St. John's Wort)
   3. CYP3A substrates with narrow therapeutic window (including, but not limited to, alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus).
8. Women who are pregnant or breastfeeding.
9. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medications.
10. Patients at risk for GI perforation.
11. Clinically significant cardiovascular disease including:

    1. QTcF interval >450 ms for men and >470 ms for women, symptomatic bradycardia <45 beats per minute or other significant ECG abnormalities in the investigator's opinion.
    2. Clinically uncontrolled hypertension in the investigator's opinion (e.g., blood pressure >160/100 mmHg; note that isolated elevated readings considered to not be indicative of uncontrolled hypertension are allowed).

    The following within 6 months prior to Cycle 1 Day 1:
    1. Congestive heart failure (New York Heart Class III or IV).
    2. Arrhythmia or conduction abnormality requiring medication. Note: patients with atrial fibrillation/flutter controlled by medication and arrhythmias controlled by pacemakers are eligible.
    3. Severe/unstable angina, coronary artery/peripheral bypass graft, or myocardial infarction.
    4. Cerebrovascular accident or transient ischemia.
12. Patients who are immunosuppressed (including known HIV infection), have a serious active infection at the time of treatment, have interstitial lung disease/pneumonitis, or have any serious underlying medical condition that would impair the ability of the patient to receive protocol treatment. Patients with controlled hepatitis C, in the investigator's opinion, are allowed. Patients with known hepatitis B must be HBeAg and HB viral DNA negative for enrollment. Note that, because of the high prevalence, all patients in the Asia-Pacific region (except Australia, New Zealand, and Japan) must be tested and, if HBsAg positive, must be HBeAg and HB viral DNA negative for enrollment.
13. Known hypersensitivity to tartrazine, a dye used in the ensartinib 100 mg capsule.
14. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
15. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the patient to be enrolled.
16. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

    Note the following pertains to patients enrolled in France
17. In France, a subject will not be eligible when under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 36 months
  as assessed by independent radiology review based on RECIST v. 1.1 criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 48 months
  Time in months from date of randomization to death due to any cause
CNS response rate | 36 months
  Based on IRR, time to CNS progression (based on IRR), objective response rate (based on IRR)
ORR based on independent radiology review | 36 months
  The proportion of patients in ITT who have an objective response (i.e., those who achieve a best response of CR or PR) per RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Selvaggi, MD, Study Chair — CEO
Locations (72):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Providence Portland Medical Center, Portland, Oregon
- Sanatorio Parque S.A., Rosario, Argentina
- Australia (3):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Chris O Brien Lifehouse, Camperdown
- Catholic University of Louvain (UCL) - Site Mont Godinne, Yvoir, Belgium
- Brazil (4):
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo
  - Hospital de Câncer de Barretos - Fundação Pio XII, São Paulo, São Paulo
  - Hospital Haroldo Juaçaba - Instituto do Cancêr do Ceará, Fortaleza
  - Fundacao do ABC Faculdade de Medicina do ABC, São Paulo
- Infirmière recherche Clinique, IUCPQ, Québec, Quebec, Canada
- China (21):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Cancer Hospital, Changsha, Hu'nan
  - Union Hospital of Tongji Medical College of Huazhong Science and Techology University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Peking University Cancer Hospital, Beijing
  - Zhejiang Cancer Hospital, Hangzhou
- Czechia (2):
  - Vítkovická Nemocnice , a.s., Ostrava-Vitkovice
  - Krajská zdravotní, a.s., Masarykova nemocnice, Ústí nad Labem
- France (4):
  - CHRU Lille, Lille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU de Rennes Hôpital Pontchaillou, Rennes
  - Hopital Saint-Louis, Vellefaux
- Germany (2):
  - Charite Campus Virchow-Klinikum, Berlin
  - Lungen Clinic Grosshansdorf, Großhansdorf
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - The University of Hong Kong/Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center Institute of Oncology, Davidoff Center, Petah Tikva
- Italy (3):
  - IEO Istituto Europeo di Oncologia, Milan
  - Centro Operativo Studi Clinici S.C.Oncologia Medica, Perugia
  - Azienda Socio Sanitaria Territoriale (ASST) della Valtellina e dell'Alto Laria, Sondrio
- Netherlands (2):
  - VU Medical Center, Amsterdam
  - Maastricht University Medical Centre (MUMC), Maastricht
- Medical University of Gdansk, Gdansk, Poland
- Russia (6):
  - Federal State Budgetary Scientific Institution Russian Oncological Scientific Center named after N.N. Blokhin, Moscow
  - LLC "Vitamed", Moscow
  - Moscow City Oncology Hospital #63, Moscow
  - BIH of Omsk Region "Clinical Oncology Dispensary", Omsk
  - Pavlov First Medical University, Saint Petersburg
  - Petrov Research Institute of Oncology, Saint Petersburg
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Son Ltatzer, Palma de Mallorca
- Trakya University Balkan Oncology Hospital, Edirne, Turkey (Türkiye)
- United Kingdom (4):
  - Blackpool Victoria Hospital, Blackwood
  - Southmead Hospital, Bristol
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Kings Mill Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horn L, Wang Z, Wu G, Poddubskaya E, Mok T, Reck M, Wakelee H, Chiappori AA, Lee DH, Breder V, Orlov S, Cicin I, Cheng Y, Liu Y, Fan Y, Whisenant JG, Zhou Y, Oertel V, Harrow K, Liang C, Mao L, Selvaggi G, Wu YL. Ensartinib vs Crizotinib for Patients With Anaplastic Lymphoma Kinase-Positive Non-Small Cell Lung Cancer: A Randomized Clinical Trial. JAMA Oncol. 2021 Nov 1;7(11):1617-1625. doi: 10.1001/jamaoncol.2021.3523. PMID 34473194